CLINICAL TRIAL: NCT01492738
Title: The Effect of Acupuncture on Anxiety and Working Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUHS H1011
Record Dates: First submitted 2011-12-01; First posted 2011-12-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Memory Impairment; Anxiety
Keywords: Acupuncture; anxiety; memory
MeSH Terms: conditions — Memory Disorders; Anxiety Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Participants will be asked to make themselves comfortable lying on a massage table for 20 minutes.
- Acupuncture group (Active Comparator): Acupuncture group will receive one acupuncture treatment for twenty minutes.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — After completing questionnaires and anxiety survey, a licensed acupuncturist will insert needles according to Clean Needle Technique into specific acupuncture points. Procedure will last 20 minutes.Following acupuncture treatment, participants will complete anxiety survey and memory test.
  Arms: Acupuncture group

SUMMARY:
This study endeavors to examine the relationship between acupuncture, anxiety, and performance on a test of working memory. In the study, all participants will complete the State-Trait Anxiety Inventory (STAI) survey to determine how anxious they are at the moment and how anxious they tend to be in general. Then ½ of subjects will receive acupuncture for 20 minutes and ½ will rest quietly for 20 minutes. After this period, all subjects will again complete the STAI survey. Then all subjects will complete the Automated Operations Span Task (AOSPAN) which is a computerized test of working memory. Statistical analysis will be performed to determine if acupuncture had any effect on State-level anxiety and on performance on the AOSPAN.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate University student
* Fluent in English
* Willing to receive acupuncture
* Aged 18-30
* In good health
* Not pregnant
* Not breastfeeding

Exclusion Criteria:

* Not an Undergraduate University student
* Not fluent in English
* Unwilling to receive acupuncture
* Under 18 years of age or older than 30 years of age
* Chronic disease
* Pregnant
* Breastfeeding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in anxiety level | Baseline and after1 hour
  Participants will complete the State-Trait Anxiety Inventory survey to see how anxious they are initially; after acupuncture treatment or quiet resting, they will complete the survey again to see how anxious they are after the intervention.
Memory task | After 1 hour
  Following acupuncture treatment or resting control, participants will complete a standardized memory test (AOSPAN) to see if intervention affects memory.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bussell, MSOM, LAc, Principal Investigator — National University of Health Sciences; Hui Yan Cai, PhD, LAc, Study Director — National University of Health Sciences
Locations (2):
- United States (2):
  - Tiffani Kim Institute, Chicago, Illinois
  - A Center for Oriental Medicine, Wilmette, Illinois